CLINICAL TRIAL: NCT06870019
Title: Effects of GPS Tracking on Patient Adherence to Hepatitis C Treatment Among People Experiencing Unsheltered Homelessness
Brief Title: Hepatitis C Tracker Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Ventura County Medical Center (Other Government)
Responsible Party: Principal Investigator, Camillo Zaks, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ISHF-62320
Record Dates: First submitted 2025-02-07; First posted 2025-03-11 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Hepatitis C Virus Infection
Keywords: Street medicine; Unsheltered homelessness; Hepatitis C; GPS tracker; Mixed-methods; Ill-housed person
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Masking Description: Masking at the participant and provider levels is not possible because participants will be randomized to receive a physical GPS tracker device or to not receive a GPS tracker device. Street medicine team providers need to know the randomization assignment to ping the tracker for scheduled medical encounters to locate the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard HCV treatment (No Intervention): Participants randomized to this study arm will receive the standard medical care for Hepatitis C.
- Standard HCV treatment + GPS tracker device (Active Comparator): Participants randomized to this study arm will receive the standard medical care for Hepatitis C and a GPS tracker device.
  Interventions: Behavioral: GPS tracker device

INTERVENTIONS:
Behavioral: GPS tracker device — GPS tracker device
  Arms: Standard HCV treatment + GPS tracker device

SUMMARY:
The goal of this study is to determine if GPS tracking can enhance adherence to hepatitis C treatment among patients diagnosed with hepatitis C infection who are also experiencing unsheltered homelessness and receiving street medicine. Research will compare medication adherence among participants randomly assigned to receive standard medical care for Hepatitis C versus the standard medical care for Hepatitis C along with GPS tracking assistance.

DETAILED DESCRIPTION:
Previous research on Hepatitis C infection (HCV) has found positivity rates between 12% and 27% among people experiencing homelessness; far exceeding typical rates found among a general housed population (1%). The usual course of HCV care in the healthcare system is screening and diagnosis in primary care, then referral to specialty care (such as Hepatology or Gastroenterology) for treatment. All of this takes place within the confines of traditional "brick and mortar" clinics. This screen, refer, and treat model presents a multitude of person- and systems-level barriers for individuals experiencing homelessness.

Street Medicine was developed as an alternative healthcare delivery model to better account for the unique circumstances of the unsheltered homeless population and better meet their healthcare needs. It is defined as the delivery of individually tailored health and social services to people experiencing unsheltered homelessness directly in their own environment. Street Medicine clinicians are ideally positioned to screen, diagnose, and treat patients for HCV. Treatment of uncomplicated HCV requires daily medication for 8 to 12 weeks. Our pilot data show that USC Street Medicine can successfully engage patients in HCV treatment on the street (93% successful follow-up rate), however, adequate longitudinal follow-up for effective treatment has been a problem for other programs.

Innovative, practical, and ethical solutions to help locate patients experiencing homelessness who require follow-up for medical treatment are needed. One such potential solution is the use of discreet GPS tracking devices that may be activated when providers are in the field to locate and provide care to patients. GPS tracking devices have been used by other Street Medicine programs caring for patients experiencing homelessness. However, no research has used GPS devices for the treatment of HCV amongst people experiencing unsheltered homelessness or formally elicited the patient perspective.

This study seeks to evaluate the impact of using a GPS tracker among patients engaged in street-based treatment for HCV on medication adherence. This is a multi-site randomized controlled study to test the impact of using a GPS tracker vs. usual care (no tracker) on HCV medication adherence, along with individual interviews to explore the perspective of unsheltered homeless patients engaged in both study arms.

In this study, the use of the GPS tracker constitutes the experimental research; not the treatment for HCV. Initial screening for HCV will have already occurred as part of usual street medicine healthcare prior to this study and will not be conducted as part of this research.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Hepatitis C infection
* Experiencing unsheltered homelessness at study initiation
* Speaks English or Spanish
* Receiving street medicine care
* Meet the American Association for the Study of Liver Diseases (AASLD) criteria for simplified treatment of Hepatitis C

Exclusion Criteria:

* Prior engagement in HCV treatment
* Decompensated cirrhosis; HBsAg positive
* Current pregnancy; Known or suspended hepatocellular carcinoma
* Prior liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence Rate | 8-12 weeks
  Number of prescribed HCV pills taken (missing from pill organizer) versus number of HCV pills prescribed (present in pill organizer) per week, for each week of the 12-week treatment regimen
Length of treatment course | 8-12 weeks
  Number of weeks patient engaged in HCV medication treatment

SECONDARY OUTCOMES:
Sustained virologic response | through study completion, an average of 24 weeks
  "Undetectable" quantitative HCV RNA blood value 12-weeks post conclusion of HCV treatment course

CONTACTS AND LOCATIONS:
Overall Officials: Camilo Zaks, MD, Principal Investigator — University of Southern California, Keck School of Medicine of USC, Department of Family Medicine, USC Street Medicine; Tipu Kahn, MD, Principal Investigator — Ventura County Medical Center
Locations (2):
- United States (2):
  - USC Street Medicine, Alhambra, California
  - Ventura County Medical Center, Ventura, California

IPD SHARING:
Plan to Share IPD: Undecided
The condition of interest for this study (HCV) is a sensitive one and thus, individual participant data will not be shared. However, de-identified data and/or data in aggregate may be shared as long as it cannot be traced back to an individual. GPS location data will not be shared; instead, data associated with the GPS device such as lost device, device used to locate participant, device refusal, etc. may be shared.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-24): https://cdn.clinicaltrials.gov/large-docs/19/NCT06870019/Prot_SAP_000.pdf